CLINICAL TRIAL: NCT02317055
Title: Magnetic Resonance Imaging Evaluation of the Tissular Oxygen Saturation in Brain
Acronym: GADOXY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment problem
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Université Joseph Fourier (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2013-A00917-38; 1321 (Other: N°sponsor)
Record Dates: First submitted 2014-12-10; First posted 2014-12-15 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Cerebral Tumor; Stroke
Keywords: MRI; Oxygenation; nirs
MeSH Terms: conditions — Stroke | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient (Other): Imaging
  Interventions: Other: imaging
- healthy subject (Other): Imaging
  Interventions: Other: imaging

INTERVENTIONS:
Other: imaging

SUMMARY:
The purpose of this study is to measure the tissular oxygen saturation in brain by magnetic resonance imaging on subjects and to correlate the results with near infrared spectroscopy measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers or Patients with cerebral lesion

Exclusion Criteria:

* claustrophobia
* MRI exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
MRI measurements of local oxygen saturation in the brain | 1 Day

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Grenoble, Grenoble, France